CLINICAL TRIAL: NCT00106184
Title: Rituximab Therapy in Refractory Adult and Juvenile Idiopathic Inflammatory Myopathy (IIM)
Brief Title: Rituximab for the Treatment of Refractory Adult and Juvenile Dermatomyositis (DM) and Adult Polymyositis (PM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Genentech, Inc. (Industry); Biogen (Industry)
Responsible Party: Principal Investigator, Chester Oddis, MD, Professor of Medicine, University of Pittsburgh, Division of Rheumatology and Clinical Immunology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N01 AR042273; 5R01AR061298-02 (NIH); HHSN26420042273C; NCT00393237 (obsolete NCT alias)
Record Dates: First submitted 2005-03-21; First posted 2005-03-22 (Estimated); Results first posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Myositis; Dermatomyositis; Polymyositis; Juvenile Dermatomyositis
Keywords: rituximab; myositis; dermatomyositis; polymyositis; refractory; Juvenile Dermatomyositis
MeSH Terms: conditions — Myositis; Dermatomyositis; Polymyositis | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Adult Study Group 1 (Experimental): Refractory adult polymyositis patients who will receive rituximab at Weeks 0 and 1 followed by placebo at Weeks 8 and 9 (Treatment Group A)
  Interventions: Drug: Rituximab; Drug: Placebo
- Adult Study Group 2 (Experimental): Refractory adult polymyositis patients who will receive placebo at Weeks 0 and 1 followed by rituximab at Weeks 8 and 9 (Treatment Group B)
  Interventions: Drug: Rituximab; Drug: Placebo
- Adult Study Group 3 (Experimental): Adult dermatomyositis patients who will receive rituximab at Weeks 0 and 1 followed by placebo at Weeks 8 and 9 (Treatment Group A)
  Interventions: Drug: Rituximab; Drug: Placebo
- Adult Study Group 4 (Experimental): Adult dermatomyositis patients who will receive placebo at Weeks 0 and 1 followed by rituximab at Weeks 8 and 9 (Treatment Group B)
  Interventions: Drug: Rituximab; Drug: Placebo
- JDM Study Group 1 (Experimental): Refractory juvenile dermatomyositis patients who will receive rituximab at Weeks 0 and 1 followed by placebo at Weeks 8 and 9 (Treatment Group A)
  Interventions: Drug: Rituximab; Drug: Placebo
- JDM Study Group 2 (Experimental): Refractory juvenile dermatomyositis patients who will receive placebo at Weeks 0 and 1 followed by rituximab at Weeks 8 and 9 (Treatment Group B)
  Interventions: Drug: Rituximab; Drug: Placebo

INTERVENTIONS:
Drug: Rituximab — Treatment Group A - intravenous rituximab 750mg/m2 BSA (Body Surface Area) up to a maximum dose of 1 gram at Weeks 0 and 1 Group B - intravenous rituximab 750mg/m2 BSA (Body Surface Area) up to a maximum does of 1 gram at Weeks 8 and 9
  Other Names: Rituxan
Drug: Placebo — Treatment Group A: placebo infusion at Weeks 8 and 9
  Treatment Group B: placebo infusion at Weeks 0 and 1

SUMMARY:
Rituximab is a man-made antibody used to treat certain types of cancer. This study will determine whether rituximab is an effective treatment for adult and pediatric patients with dermatomyositis or polymyositis.

Study hypotheses: 1) The time to improvement in Group A patients (receiving rituximab first) will occur significantly earlier than in Group B patients (receiving rituximab later). 2) The proportion of patients improved at Week 8 of the treatment phase will be significantly greater in Group A than in Group B.

DETAILED DESCRIPTION:
Rituximab is a chimeric, murine-human, genetically engineered monoclonal antibody directed against the CD20 (cluster of differentiation antigen 20) antigen found on the surface of B-lymphocytes and is known to deplete B cells when administered intravenously. It is approved to treat non-Hodgkin's lymphoma. Rituximab has been used for autoimmune diseases such as systemic lupus erythematosus (SLE), rheumatoid arthritis (RA), and immune-mediated hematologic disorders. It has also been studied and used in small numbers of patients with myositis. This study will evaluate the efficacy of rituximab in treating refractory adult and pediatric patients with dermatomyositis and adult polymyositis.

A patient's participation in this study will last approximately 45 weeks. At screening, participants will have a physical exam, muscle strength assessment, an electrocardiogram, and blood and urine collection; they will also be asked to complete several questionnaires. All participants will receive 2 infusions of rituximab and 2 infusions of placebo. Participants will be randomly assigned to one of two groups. Group A will receive rituximab at Weeks 0 and 1 and placebo at Weeks 8 and 9. Group B will receive placebo at Weeks 0 and 1 and rituximab at Weeks 8 and 9. Each infusion will be given on an outpatient basis over a minimum of approximately 5 hours' time.

There will be a total of 14 study visits. All participants will visit the outpatient clinic at selected time points for muscle strength testing, a physical exam, disease activity measurements, and blood collection. During the study, participants will be monitored closely for improvement or worsening of their disease and for serious drug related side effects. Some participants will be asked if they are willing to undergo 2 muscle biopsy procedures, 1 prior to receiving study medication and 1 after receiving study medication, to determine the effects of rituximab on muscle tissue.

If a participant is unable to locate a near-by clinical center, the adult and pediatric centers at the National Institute of Health located in Bethesda, Maryland have funds available to assist with travel costs.

NIH SUB-STUDY: "Rituximab to Treat Dermatomyositis and Polymyositis"

* This study is currently recruiting patients.
* Sponsored by: National Institute of Environmental Health Sciences (NIEHS)
* Information provided by: National Institutes of Health Clinical Center (CC)
* Expected Total Enrollment: 30
* Study start: October 2006
* Location and Contact Information: Patient Recruitment and Public Liaison Office;(800) 411-1222; prpl@mail.cc.nih.gov; Phone: 1-866-411-1010

The NIH sub-study will take advantage of the multi-center core RIM trial to identify changes in gene expression patterns in muscle, skin, and peripheral blood and the imaging features and immunopathology of muscle, skin, and peripheral cells before (week 0) and after (week 16) therapy. These changes will also be correlated with the large number of clinical, laboratory, and research variables already planned to be collected in the core RIM Study. Furthermore, knowing specifically which gene expression patterns are altered in resistant patients before rituximab, and which are changed after rituximab therapy - in conjunction with flow cytometry of peripheral cells and immunopathology of the tissues - will help in understanding more about the pathogenesis of myositis and the possible contribution of B lymphocytes and their subsets.

Patients with dermatomyositis and polymyositis who meet the inclusion/exclusion criteria for the core RIM trial may be eligible for this sub-study. The following procedures will be conducted in addition to the core RIM trial procedures during the 13 clinic visits over a period of 44 weeks:

* Weeks 0, 16: Muscle and skin biopsy (adult only). Small samples of muscle and skin tissue will be surgically removed for examination under a microscope.
* Weeks 0, 8, 16, 44: Skin evaluation and photography. The effect of the disease on the skin will be thoroughly evaluated and photographs of any rashes and of the skin around the nails will be taken.
* Weeks 0, 8, 16, 44: Magnetic resonance imaging (MRI). All participants will have MRI scans of the skin and of the muscle in the legs. Adults will also have an MRI to examine blood flow in the muscle.

ELIGIBILITY:
Inclusion Criteria:

* Adults with definite or probable dermatomyositis or polymyositis and pediatric patients five years of age and over with definite or probable juvenile dermatomyositis (JDM) by Bohan and Peter criteria. Diagnosis of JDM based on an age of onset (i.e., first symptom of myositis or dermatomyositis rash) is less 18 years of age
* Refractory myositis, defined by intolerance to or inadequate response to corticosteroids plus an adequate regime of at least one other immunosuppressive agent. Intolerance is defined as side effects that require discontinuation of the medication or an underlying condition that precludes further use of the medication.
* Baseline manual muscle testing which is based on a maximum MMT-8 (Manual Muscle Test) score of 150:Adult subjects with dermatomyositis (DM) or polymyositis (PM) must have a score that is no greater than 125/150 in conjunction with 2 other abnormal core set measures.

Subjects with a diagnosis of Juvenile Dermatomyositis (JDM) must meet either of the following criteria:

1. An MMT-8 (Manual Muscle Test) score that is no greater than 125/150 in conjunction with 2 other abnormal core set measures.

   OR
2. If MMT (Manual Muscle Test) score is greater than 125/150 the patient MUST meet at least 3 abnormal core set measures.

   * Background therapy with at least 1 non-corticosteroid immunosuppressive agent at a stable dose for at least 6 weeks prior to screening
   * Able and willing to complete self-report questionnaires. Parents of pediatric participants will be required to complete the questionnaires on behalf of their children.
   * Willing to use acceptable forms of contraception for the duration of the study for patients of reproductive potential.
   * Parent willing to provide informed consent, if applicable
   * Willing to forgo immunization with a live vaccine for the duration of the study

Exclusion Criteria:

* Drug-induced myositis. Patients who have myositis or myopathic syndromes caused by taking medications known to induce myositis-like syndromes, including but not limited to statin agents, fibric acid derivatives, colchicine, and hydroxychloroquine.
* Juvenile polymyositis
* Inclusion body myositis
* Cancer-associated myositis, defined as the diagnosis of myositis within 2 years of the diagnosis of cancer. Patients with basal or squamous cell skin cancer or carcinoma in situ of the cervix are not excluded, if it has been at least 5 years since excision.
* Myositis in overlap with another connective tissue disease that may preclude the accurate assessment of a treatment response
* Live viral vaccine within 4 weeks prior to study entry
* Any joint disease or other musculoskeletal condition that may interfere with muscle strength testing
* Known hypersensitivity to mouse proteins
* Any concomitant or life-threatening non-myositis illness that, in the opinion of the investigator, may interfere with the study
* Known or suspected history of drug or alcohol abuse within the last 6 months prior to study entry, as determined by medical record or patient interview
* Anticipated poor compliance with study requirements
* Participation in another clinical trial within 30 days prior to screening
* Any history or evidence of any severe illness or other condition that, in the opinion of the investigator, may interfere with the study
* Previously received rituximab
* Evidence of prior infection with hepatitis B or hepatitis C virus
* Initiation of an exercise program within 4 weeks of screening OR initiation of an exercise program during the study
* Consumed any creatine-containing, over-the-counter products in the form of dietary supplements 30 days prior to screening visit and for the duration of the study

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-03; Primary Completion 2010-02 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chester V. Oddis, MD, Principal Investigator — University of Pittsburgh; Ann M. Reed, MD, Principal Investigator — Mayo Clinic
Locations (31):
- United States (27):
  - University of Alabama Arthritis Intervention Program (Adult Site), Birmingham, Alabama
  - Phoenix Neurological Associates, LTD (Adult Site), Phoenix, Arizona
  - Cedars-Sinai Medical Center (Adult Site), Los Angeles, California
  - Stanford University (Adult Site), Stanford, California
  - Stanford University (Pediatric Site), Stanford, California
  - University of Miami School of Medicine (Adult Site), Miami, Florida
  - Miami Children's Hospital (Pediatric Site), Miami, Florida
  - University of Kansas Medical Center (Adult Site), Kansas City, Kansas
  - Kentucky Clinic (Adult Site), Lexington, Kentucky
  - National Institute of Health (Adult Site), Bethesda, Maryland
  - National Institute of Health (Pediatric Site), Bethesda, Maryland
  - Children's Hospital of Boston (Pediatric Site), Boston, Massachusetts
  - Beth Israel Deaconess Medical Center (Adult Site), Boston, Massachusetts
  - University of Michigan Health System (Adult Site), Ann Arbor, Michigan
  - Michigan State University (Adult and Pediatric Site), Grand Rapids, Michigan
  - Mayo Clinic (Adult Site), Rochester, Minnesota
  - Mayo Clinic (Pediatric Site), Rochester, Minnesota
  - North Shore Long Island Jewish Health System (Adult Site), Lake Success, New York
  - Hospital for Special Surgery (Adult Site), New York, New York
  - Duke University Medical Center (Pediatric Site), Durham, North Carolina
  - Cincinnati's Children's Hospital (Pediatric Site), Cincinnati, Ohio
  - Children's Hospital of Philadelphia (Pediatric Site), Philadelphia, Pennsylvania
  - University of Pennsylvania (Adult Site), Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh (Pediatric Site), Pittsburgh, Pennsylvania
  - University of Pittsburgh / UPMC (Adult Site), Pittsburgh, Pennsylvania
  - University of Texas Southwestern Medical Center (Adult), Dallas, Texas
  - Medical College of Wisconsin / Froedtert Memorial Luthern Hospital (Adult Site), Milwaukee, Wisconsin
- Canada (2):
  - IWK Health Centre, Halifax, Nova Scotia
  - Hospital for Sick Children (Pediatric Site), Toronto, Ontario
- Institute of Rheumatology, Prague, Czechia
- Karolinska Institute, Stockholm, Sweden

REFERENCES:
- [Background] Feldman B, Wang E, Willan A, Szalai JP. The randomized placebo-phase design for clinical trials. J Clin Epidemiol. 2001 Jun;54(6):550-7. doi: 10.1016/s0895-4356(00)00357-7. PMID 11377114
- [Background] Levine TD. Rituximab in the treatment of dermatomyositis: an open-label pilot study. Arthritis Rheum. 2005 Feb;52(2):601-7. doi: 10.1002/art.20849. PMID 15692974
- [Result] Oddis CV, Reed AM, Aggarwal R, Rider LG, Ascherman DP, Levesque MC, Barohn RJ, Feldman BM, Harris-Love MO, Koontz DC, Fertig N, Kelley SS, Pryber SL, Miller FW, Rockette HE; RIM Study Group. Rituximab in the treatment of refractory adult and juvenile dermatomyositis and adult polymyositis: a randomized, placebo-phase trial. Arthritis Rheum. 2013 Feb;65(2):314-24. doi: 10.1002/art.37754. PMID 23124935
- See also: Click here for the Myositis Association Web site — http://www.myositis.org
- See also: Click here for the NIH Clinical Center (sub-study) — http://clinicalstudies.info.nih.gov/cgi/wais/bold032001.pl?A_07-E-0012.html@myositis

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject were screened and enrolled at 26 US and 4 international sites.
Pre-assignment Details: In an effort to exclude IBM (Inclusion Body Myositis) and other myositis mimics, the medical records and muscle biopsy results (if available) of adults with PM were reviewed by a 3-member Adjudication Committee before enrollment.
Groups:
- Treatment Group A (Rituximab Wks 0 and 1): Subjects received rituximab at Weeks 0 and 1 followed by placebo at Weeks 8 and 9 (Treatment Group A)
  Rituximab : Treatment Group A - intravenous rituximab 750mg/m2 BSA (Body Surface Area) up to a maximum dose of 1 gram at Weeks 0 and 1 Placebo : Treatment Group A: placebo infusion at Weeks 8 and 9
- Treatment Group B (Rituximab Wks 8 and 9): Subjects received placebo at Weeks 0 and 1 followed by rituximab at Weeks 8 and 9 (Treatment Group B)
  Group B - intravenous rituximab 750mg/m2 BSA up to a maximum does of 1 gram at Weeks 8 and 9
  Treatment Group B: placebo infusion at Weeks 0 and 1
Period: Overall Study
Arm/Group | Treatment Group A (Rituximab Wks 0 and 1) | Treatment Group B (Rituximab Wks 8 and 9)
Started | 96 | 104
Treated | 93 (96 subjects were randomized.) | 102 (104 subjects were randomized.)
Completed | 93 | 102
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: 3 subjects in Group A and 2 subjects in Group B were excluded from analysis due to withdrawing from the study. These subjects either did not receive a full dose of study drug at week 0 or no study drug at all.
Groups:
- Group A: Subjects received rituximab at Weeks 0 and 1 followed by placebo at Weeks 8 and 9 (Treatment Group A)
  Rituximab : Treatment Group A - intravenous rituximab 750mg/m2 BSA up to a maximum dose of 1 gram at Weeks 0 and 1
  Placebo : Treatment Group A: placebo infusion at Weeks 8 and 9
- Group B: Subjects received placebo at Weeks 0 and 1 followed by rituximab at Weeks 8 and 9 (Treatment Group B)
  Group B - intravenous rituximab 750mg/m2 BSA up to a maximum does of 1 gram at Weeks 8 and 9
  Treatment Group B: placebo infusion at Weeks 0 and 1
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 96 | 104 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 19 | 36
  Between 18 and 65 years | 70 | 80 | 150
  >=65 years | 9 | 5 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (18.23) | 40.7 (18.4) | 41.8 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 78 | 146
  Male | 28 | 26 | 54
Region of Enrollment [Number; unit: participants]
  United States | 87 | 98 | 185
  Czech Republic | 4 | 3 | 7
  Canada | 2 | 3 | 5
  Sweden | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Comparison Between the Time to Improvement Between the Two Groups of IIM (Idiopathic Inflammatory Myopathy) Patients
Description: The Definition of Improvement for both adult and pediatric patients will be: 3 of any of the 6 core set measures improved by ≥ 20%, with no more than 2 of the core set measures worsening by ≥25% (worsening measure cannot include the MMT) at two consecutive visits. Of note, the MMT could not be one of the worsening measures.
  Core Set Measures Included:
  1. Manual Muscle Testing (MMT)- Muscle Strength
  2. Physician Global Disease Activity VAS Score
  3. Health Assessment Questionnaire Index Score - Physical Function
  4. Patient Global Assessment of Disease Activity VAS score
  5. Extramuscular Activity - Myositis Disease Activity Assessment Tool
  6. 2 or more elevated muscle enzymes (Aldolase, CK, AST, ALT, and LDH)
Time Frame: Week 44 of treatment phase
Population: Intention to Treat (ITT)
Measure: Median (Full Range); unit: Weeks
Groups:
- Group A (Rituximab Wks 0 and 1): Subjects received rituximab at Weeks 0 and 1 followed by placebo at Weeks 8 and 9 (Treatment Group A)
  Rituximab : Treatment Group A - intravenous rituximab 750mg/m2 BSA up to a maximum dose of 1 gram at Weeks 0 and 1
  Placebo : Treatment Group A: placebo infusion at Weeks 8 and 9
- Group B (Rituximab Wks 8 and 9): Group B - intravenous rituximab 750mg/m2 BSA up to a maximum does of 1 gram at Weeks 8 and 9
  Treatment Group B: placebo infusion at Weeks 0 and 1
Arm/Group | Group A (Rituximab Wks 0 and 1) | Group B (Rituximab Wks 8 and 9)
Number analyzed (Participants) | 96 | 104
Weeks | 20.2 [8 to 44] | 20.0 [8 to 44]
Statistical Analysis 1: Comparison: Group A (Rituximab Wks 0 and 1) vs Group B (Rituximab Wks 8 and 9); Proportional hazards model; Test type: Superiority or Other; p = 0.74, Log Rank; No confidence intervals as no parameters were estimated

2. Secondary Outcome: Response Rates (Proportion of Improved Patients) Between Groups A (Rituximab Wks 0 and 1) and B (Rituximab Wks 8 and 9) at Week 8
Description: as for outcome 1
Time Frame: Week 8 of the treatment phase
Population: Intention to Treat (ITT)
Measure: Number; unit: participants
Groups:
- Treatment Group A (Rituximab Wks 0 and 1): Subjects received rituximab at Weeks 0 and 1 followed by placebo at Weeks 8 and 9 (Treatment Group A)
  Rituximab : Treatment Group A - intravenous rituximab 750mg/m2 BSA up to a maximum dose of 1 gram at Weeks 0 and 1 Placebo : Treatment Group A: placebo infusion at Weeks 8 and 9
Arm/Group | Treatment Group A (Rituximab Wks 0 and 1) | Treatment Group B (Rituximab Wks 8 and 9)
Number analyzed (Participants) | 96 | 104
participants | 14 | 21
Statistical Analysis 1: Comparison: Treatment Group A (Rituximab Wks 0 and 1) vs Treatment Group B (Rituximab Wks 8 and 9); Test type: Superiority or Other; p > 0.90, Chi-squared; Difference in baseline muscle enzymes therefore tested the difference in the proportions adjusting for the baseline values

3. Secondary Outcome: 20% Improvement in Manual Muscle Testing (MMT) Over Baseline on Two Consecutive Time Points (Muscle is the Primary Organ of Involvement, and MMT is the One Objective Measurement of the Definition of Improvement [DOI])
Description: Number of participants with a 20% improvement in MMT over baseline on two consecutive time points.
Time Frame: Week 44 of treatment phase
Population: Intention to Treat (ITT)
Measure: Number; unit: Participants
Arm/Group | Treatment Group A (Rituximab Wks 0 and 1) | Treatment Group B (Rituximab Wks 8 and 9)
Number analyzed (Participants) | 96 | 104
Participants | 14 | 21
Statistical Analysis 1: Comparison: Treatment Group A (Rituximab Wks 0 and 1) vs Treatment Group B (Rituximab Wks 8 and 9); Test type: Superiority or Other; p > 0.90, Log Rank

ADVERSE EVENTS:
Time Frame: Reported Adverse Events (AEs) include events starting on or after Week 0 and on or before Week 44 of the study.
Groups:
- Treatment Group A: Subjects received rituximab at Weeks 0 and 1 followed by placebo at Weeks 8 and 9 (Treatment Group A)
  Rituximab : Treatment Group A - intravenous rituximab 750mg/m2 BSA up to a maximum dose of 1 gram at Weeks 0 and 1 Placebo : Treatment Group A: placebo infusion at Weeks 8 and 9
- Treatment Group B: Subjects received placebo at Weeks 0 and 1 followed by rituximab at Weeks 8 and 9 (Treatment Group B)
  Group B - intravenous rituximab 750mg/m2 BSA up to a maximum does of 1 gram at Weeks 8 and 9
  Treatment Group B: placebo infusion at Weeks 0 and 1
Arm/Group | Treatment Group A | Treatment Group B
Serious Adverse Events (participants affected / at risk) | 24/96 | 41/104
Other Adverse Events (participants affected / at risk) | 45/96 | 55/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group A (N=96) | Treatment Group B (N=104)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Anemia die to esophageal ulcers
Cardiac Ischemia/myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 1 (1)
Myocarditis (Cardiac disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 2 (2) | 2 (2)
Clostridium Infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 0 (0) | 2 (2)
Histoplasmosis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 4 (4)
Raynaud Ulcer (Vascular disorders) | 1 (1) | 1 (1)
Viral Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Muscle Weakness - Disease Flare (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Infection (Infections and infestations) | 1 (1) | 0 (0)
Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Neurological Disorder - Aseptic Meningitis (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Kidney Stones (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Surgical Procedure (Surgical and medical procedures) | 1 (1) | 7 (7)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Death - Cerebral Vascular Accident (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group A (N=96) | Treatment Group B (N=104)
Headache (General disorders) | 13 (13) | 12 (12)
Nausea (Gastrointestinal disorders) | 10 (10) | 10 (10)
Bronchitis (Infections and infestations) | 6 (6) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 9 (9)
Fever (General disorders) | 6 (6) | 10 (10)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 10 (10)

LIMITATIONS AND CAVEATS:
There was an overestimate of the rapidity of the rituximab response and an underestimate of DOI in those receiving placebo.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No